CLINICAL TRIAL: NCT01627119
Title: The Functional and Clinicopathological Roles and Therapeutic Implication of Connective Tissue Growth Factor in Peritoneal Metastasis of Gastric Cancer
Acronym: CTGF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, MD, PhD, National Taiwan University Hospital
Other Study IDs: 200906054R
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Gastric Cancer
Keywords: CTGF; Peritoneal metastasis
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Cancer tissue and adjacent normal tissue Urine Blood serum and blood plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Gastric cancer patients: Gastric cancer patients who receive curative surgery at National Taiwan University Hospital

SUMMARY:
For the past 50 years, gastric cancer has been one of the ten most frequent cancers and the second leading cause of cancer-related death in the world. In Taiwan, it is the fifth most common cause of cancer-related deaths, accounting for 6.3% of all cancer deaths. The poor prognosis of gastric cancer is mostly caused by the extensive metastasis to the lymph nodes, liver, and peritoneal dissemination even if curative resection was performed. The main cause of recurrence after curative or noncurative resection of advanced tumors is peritoneal metastasis because of possible direct spillage and dissemination of tumor cells as a result of surgical manipulation, and it is associated with a poor prognosis. As yet, no effective treatment has been developed for this condition. The development of peritoneal metastasis is a multistep process, beginning with attachment to peritoneal mesothelial cells, retraction of the mesothelial cells and exposure of the basement membrane, attachment to the basement membrane, degradation in the extracellular matrix, proliferation by the cancer cells, and angiogenesis, and it is clear that many types of agents are involved at the various stages of this process. Developing a new therapeutic method for this mode of metastasis is very important for improvement of gastric cancer treatment.

CTGF is a secretory protein belonging to the CCN family (one among the three originally discovered members: cysteine-rich61, CTGF, and nephroblastoma-overexpressed gene). It is a multifunctional growth factor involved in wound healing, inflammation, cell adhesion, chemotaxis, apoptosis, tumor growth, and fibrosis. Recent studies showed that overexpression of CTGF in human oral squamous cell carcinoma reduces cell growth and tumorigenecity. Similar tumor growth inhibitory effects were observed in lung cancer cells in which CTGF overexpression was less angiogenic and metastatic due to blocking of the VEGF A signaling pathway. CTGF was also reported to be a key regulator of colorectal cancer invasion and metastasis, and it appears to be a better prognostic factor. These studies suggest that CTGF may involve the processes of peritoneal metastasis which includes cancer cell adhesion in peritoneum, proliferation and angiogenesis. Peritoneal mesothelium is the first surface encountered by disseminated tumor cells and successful adhesion is, therefore, of paramount importance in metastasis formation. Therefore, we hypothesized that CTGF is a potential molecule target, which may be related to cell adhesion to peritoneum, the first step of peritoneal metastasis, and its exact mechanism may includes proliferation and angiogenesis.

In order to answer these important questions, first, we have performed the preliminary studies to prove CTGF did express in different gastric cancer cell lines including AGS, N87, TSGH, and MKN-45 by using RT-PCR and Western blotting, and gastric cancer tissues by using immunohistochemical method. Second, we demonstrated different levels of CTGF expression in different cell lines pose different adhesion ability in in-vitro adhesion assay. Third, we conducted a transient CTGF-overexpressed MKN45 gastric cancer cell line, and CTGF-overexpressed cell line had lower adhesive ability compared to the control.

Next step in this project, we will be studying the roles of CTGF plays in cellular and molecular biology in vitro and in vivo and clinical significance associated with therapeutic potential of peritoneal metastasis from gastric cancer. We will generate stable clones of MKN45 cells harboring CTGF and its control cell line to elucidate the roles of CTGF in cancer cell adhesion, proliferation and angiogenesis in peritoneum.

ELIGIBILITY:
Inclusion Criteria:

* Gastric cancer patients who are elegible for curative surgery
* Age 25-90

Exclusion Criteria:

* Gastric cancer patients who are not elegible for curative surgery

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients Age 25-90
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
To measure the expression level of CTGF in patient blood and tissue | 1 day
  To determine the level of CTGF expression in gastric cancer patient specimens collected during surgery.

SECONDARY OUTCOMES:
To determine the survival probability of gastric cancer patients after surgery | 10 years from date of surgery
  To determine the survival probability of gastric cancer patients after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chiung-Nien Chen, MD, PhD, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan